CLINICAL TRIAL: NCT07017426
Title: Fuzheng Huayu Tablets Reduce the Occurrence of Re-Decompensation Events in Patients With First Decompensation of Hepatitis B-Related Liver Cirrhosis: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study
Acronym: FZHYRORDFDHBLC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhiyun Yang (Other)
Responsible Party: Sponsor-Investigator, Zhiyun Yang, Vice President of Beijing Ditan Hospital Affiliated to Capital Medical University Affiliation: Beijing Ditan Hospital, Beijing Ditan Hospital
Organization: Beijing Ditan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BJDHYZYFZHY
Record Dates: First submitted 2025-06-05; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Decompensated Hepatitis B Cirrhosis
MeSH Terms: interventions — fuzheng huayu

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fuzheng Huayu tablets combined with conventional antiviral therapy (Experimental)
  Interventions: Drug: Fuzheng Huayu tablets
- placebo combined with conventional antiviral therapy (Placebo Comparator)
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Drug: Fuzheng Huayu tablets — Fuzheng Huayu Tablets are composed of various medicinal ingredients such as Salvia miltiorrhiza, Prunus persica seed, Gynostemma pentaphyllum, pine pollen, Cordyceps sinensis, and Schisandra chinensis. They have the functions of promoting blood circulation and removing blood stasis, nourishing the liver and enriching essence, and can be used to treat chronic liver diseases, anti-fibrosis, and patients with liver cirrhosis.
  Arms: Fuzheng Huayu tablets combined with conventional antiviral therapy
Other: Placebo Comparator — placebo combined with conventional antiviral therapy
  Arms: placebo combined with conventional antiviral therapy

SUMMARY:
This study aims to conduct a prospective, multicenter, double-blind, randomized, placebo-controlled trial. The planned sample size is 432 patients, with the ratio of the Fuzheng Huayu group to the placebo control group being 1:1. Participants will be randomly assigned to the two groups using a stratified block randomization method at the central level. The Fuzheng Huayu group (Fuzheng Huayu tablets combined with conventional antiviral therapy) and the placebo group (placebo combined with conventional antiviral therapy) will be treated for 48 weeks, followed by a 96-week follow-up. The study period will last for a total of 2 years. The cumulative incidence of recurrent decompensation events within 1 year, the cumulative incidence of recompensation within 1 year, the incidence of liver failure, liver cancer, and liver disease-related deaths will be analyzed. The efficacy and safety of Fuzheng Huayu tablets in reducing the recurrence of decompensation events in patients with first-time decompensated hepatitis B cirrhosis will be clarified, providing a basis for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily joining the group, able to understand and sign informed consent forms;
* Age range: 18-80 years old, gender not limited;
* HBsAg positive for ≥ 6 months during screening;
* Complies with traditional Chinese medicine syndrome types: blood stasis obstructing collaterals, liver and kidney deficiency syndrome;
* The first decompensated event, which meets the diagnostic criteria for decompensated cirrhosis in the "Diagnosis and Treatment Guidelines for Cirrhosis (2019 Edition)": (1) having diagnostic evidence for cirrhosis; (2) Complications related to portal hypertension may occur, such as ascites, esophageal and gastric variceal bleeding, hepatic encephalopathy, hepatorenal syndrome, etc.

Exclusion Criteria:

* Merge hepatitis A, C, D, E, and/or HIV infections;
* Merge autoimmune liver disease, alcoholic liver disease, drug-induced liver disease and other liver diseases;
* Patients with combined malignant tumors;
* History of splenectomy and transjugular intrahepatic portosystemic shunt surgery;
* Individuals with neurological and psychiatric disorders, especially those with a history of depression, anxiety, mania, schizophrenia, or a family history of mental illness (especially those with a history of depression or tendencies towards depression);
* Individuals with severe heart, lung, kidney and other organ disorders;
* Individuals who plan to undergo organ transplantation or have already undergone organ transplantation;
* Pregnant or lactating women or those with fertility plans during the study period;
* For those who are allergic to tonifying the body and removing blood stasis, nucleoside (acid) analogues, or drugs, or who meet any contraindications in the research drug instructions;
* Individuals who have taken traditional Chinese medicine such as Fuzheng Huayu within the past 6 months;
* Other situations that have participated in other intervention studies within the previous 3 months or are deemed unsuitable for inclusion by the researchers;
* The population diagnosed with liver cancer 3 months after enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
the cumulative incidence of recurrent decompensation events | 1 year

SECONDARY OUTCOMES:
the cumulative incidence of recompensation | 1 year
the incidence of liver failure | 1 year and 2 year
the incidence of liver cancer | 1 year and 2 year
the incidence of liver disease-related deaths | 1 year and 2 year